CLINICAL TRIAL: NCT00003687
Title: A Phase III Double-Blind Equivalence Study of Two Different Formulations of Slow-Release Morphine Followed by a Randomization Between Dextromethorphan or Placebo Plus Statex SR for Chronic Cancer Pain Relief in Terminally Ill Patients
Brief Title: Treatment for Chronic Pain in Patients With Advanced Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SC17; CAN-NCIC-SC17 (Other: PDQ); CDR0000066789 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Pain; Precancerous/Nonmalignant Condition; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; small intestine lymphoma; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; pain; prolymphocytic leukemia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; primary systemic amyloidosis; non-Hodgkin lymphoma during pregnancy; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; chronic eosinophilic leukemia; chronic neutrophilic leukemia; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Pain; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Lymphoma, B-Cell, Marginal Zone | interventions — Dextromethorphan; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: dextromethorphan hydrobromide
Drug: morphine sulfate

SUMMARY:
RATIONALE: Different drug formulations and combinations of drugs may help patients with chronic pain live more comfortably. It is not yet known which regimen is most effective for chronic pain.

PURPOSE: Randomized phase III trial to compare the effectiveness of different morphine formulations with or without dextromethorphan in treating chronic pain in patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the analgesic efficacy of two formulations of morphine (Statex SR versus MS-Contin) in patients requiring morphine for the treatment of chronic cancer pain.
* Compare the effect of these 2 formulations of morphine on the total analgesic consumption, sleep disturbances, sleep and nausea, responses of different types of pain, and toxic effects experienced in the two treatment groups.
* Compare the effect of coadministration of morphine and dextromethorphan versus morphine and placebo on pain control in the respective patient groups (phase B).
* Compare the effect of morphine and dextromethorphan or placebo on total analgesic consumption, sleep disturbances, sleep and nausea, responses of different types of pain, and toxic effects on the two treatment groups (phase B).

OUTLINE: This is a randomized, double-blind, parallel-group, multicenter study. Patients are stratified by stabilization dose (less than 120 mg/day vs greater than 120 mg/day of morphine) and institution in phase A, and neuropathic pain (yes vs no) in phase B.

* Phase A: Patients are randomized to receive oral morphine in one of two formulations (MS Contin or Statex SR) every 12 hours for 7 days.
* Phase B: Eligible patients from phase A who have taken no more than 2 breakthrough doses of analgesic per day in the previous 2 days are re-randomized to receive dose escalated oral dextromethorphan capsules or placebo every 4 hours, and oral morphine tablets every 12 hours for 14 days.
* Phase C: All patients fulfilling entry criteria at the end of phase A or any time during phase B may receive compassionate use morphine tablets for up to 90 days.

Patients complete a pain diary twice each day during treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven advanced cancer with chronic pain
* Cancer pain requiring strong opioids having an average pain score of less than 6/10 on the visual analog scale within last 24 hours
* Pain managed by a stable maintenance dose of MS-Contin formulation of morphine for at least 2 days with no more than 2 breakthrough immediate release morphine doses per 24 hours
* Pain that is expected to be controlled by a stable and adequate total daily dose of sustained release morphine for the first 7 days of the study

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Not specified

Life expectancy:

* At least 2 months

Hematopoietic:

* Not specified

Hepatic:

* SGOT or SGPT no greater than 3 times upper limit of normal (ULN)
* No liver disease

Renal:

* Creatinine no greater than 2 times ULN
* No kidney failure

Pulmonary:

* No clinically significant respiratory depression
* No severe obstructive airway disease

Other:

* Fluent in English or French
* No known hypersensitivity or allergy to study medications or components or other multiple drug allergies
* Normal cognition defined by the Folstein Mini-Mental State Questionnaire (at least 24/30 correct)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 14 days since prior chemotherapy

Endocrine therapy:

* Concurrent steroids allowed

Radiotherapy:

* At least 14 days since prior analgesic radiotherapy

Surgery:

* Not specified

Other:

* At least 3 months since prior investigational agents
* At least 1 month since prior clinical study
* No concurrent analgesics other than morphine
* No other concurrent medications containing dextromethorphan
* Concurrent antidepressant medication allowed
* Concurrent nonsteroidal antiinflammatory drugs allowed
* At least 14 days since prior monoamine oxidase (MAO) inhibitors
* No concurrent MAO inhibitors

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 1998-06-11 (Actual); Primary Completion 2001-09-26 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Study Chair — M.D. Anderson Cancer Center
Locations (4):
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] MacDonald S, Dudgeon DJ, Bruera E, et al.: A phase III double-blind equivalence study of two different formulations of slow-release morphine followed by a randomization between dextromethorphan or placebo plus Statex SR for chronic cancer pain relief in terminally ill patients. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1521, 2002.
- [Result] Dudgeon DJ, Bruera E, Gagnon B, Watanabe SM, Allan SJ, Warr DG, MacDonald SM, Savage C, Tu D, Pater JL. A phase III randomized, double-blind, placebo-controlled study evaluating dextromethorphan plus slow-release morphine for chronic cancer pain relief in terminally ill patients. J Pain Symptom Manage. 2007 Apr;33(4):365-71. doi: 10.1016/j.jpainsymman.2006.09.017. PMID 17397698